CLINICAL TRIAL: NCT03184311
Title: High-intensity Interval Training as Treatment Strategy for Heart Failure Patients With Preserved Ejection Fraction: A Prospective, Single-blind, Randomized Controlled Trial
Brief Title: High-intensity Interval Training in Heart Failure Patients With Preserved Ejection Fraction
Acronym: HIT-HF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Basel (Other)
Collaborators: Clinical Trial Unit, University Hospital Basel, Switzerland (Other)
Responsible Party: Principal Investigator, Arno Schmidt-Trucksäss, Clinical Director, University of Basel
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019-00188
Record Dates: First submitted 2017-06-02; First posted 2017-06-12 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Heart Failure With Normal Ejection Fraction
Keywords: Therapy response prediction; Exercise tolerance; High-intensity interval training
MeSH Terms: interventions — High-Intensity Interval Training

STUDY DESIGN:
Intervention Model Description: * Intervention group: 12-week high-intensity interval training on a bicycle ergometer.
  * Control group: 12-week moderate-intensity continuous training on a bicycle ergometer.
Who Masked: Outcomes Assessor
Masking Description: Study personnel involved in the study measurements will be blinded to whether patients are allocated to the intervention or control group. Furthermore, the statistician will be blinded to treatment allocation. To ensure blinding, the study measurements will be performed in different rooms and by different staff than those involved in the training intervention. It is not possible to blind participating patients and investigators performing the randomization and training sessions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-intensity interval training (HIT) (Experimental): A 12-week HIT will be performed 3 times per week on a bicycle ergometer according to the protocol of Wisløff et al. In the first 4 weeks of the program, all sessions will consist of moderate continuous training (MCT) at 60-80% of peak heart rate (HRpeak) for 40 minutes in order that patients get used to exercising. For weeks 4-12, the following HIT protocol is intended: Patients will warm up for 10 minutes at moderate intensity (60-70% of HRpeak, Borg 11-13) before cycling four 4-minute intervals at high intensity (85-95% of HRpeak, Borg 15-17). Each interval will be separated by a 3-minute active pause at 60-70% of HRpeak (Borg 11-13). The training session will end with a 5-minute cool-down at moderate intensity (60-70% of HRpeak). Total exercise time will be 40 minutes.
  Interventions: Other: High-intensity interval training (HIT)
- Moderate-intensity continuous training (MCT) (Placebo Comparator): A 12-week MCT will be performed 3 times per week on a bicycle ergometer. All sessions will consist of moderate continuous training (MCT) at 60-70% of peak heart rate (HRpeak) for 47 minutes.
  Interventions: Other: Moderate-intensity contiuous training (MCT)

INTERVENTIONS:
Other: High-intensity interval training (HIT) — Supervised 12-week HIT 3 times per week on a bicycle ergometer.
  Arms: High-intensity interval training (HIT)
Other: Moderate-intensity contiuous training (MCT) — Supervised 12-week MCT 3 times per week on a bicycle ergometer.
  Arms: Moderate-intensity continuous training (MCT)

SUMMARY:
This study investigates the effects of a 12-week high-intensity interval training (HIT) on exercise tolerance, functional status and quality of life in patients with chronic heart failure with preserved ejection fraction (HFpEF), in comparison to a control group undergoing a 12-week moderate-intensity continuous training.

DETAILED DESCRIPTION:
Heart failure (HF) with preserved ejection fraction (HFpEF) occurs in about 50% of all HF patients. Remodeling and fibrosis stimulated by inflammation appear to be main factors for the progression of HFpEF. The lack of prognostic treatment options in HFpEF urgently calls for new therapeutic approaches. While beneficial effects of exercise training have been demonstrated in HF with reduced ejection fraction, they have not yet been evaluated in HFpEF. Therefore, the aim of this study is to investigate the effects of high-intensity interval training (HIT) in HFpEF patients.

The proposed study will be a prospective, single-blind, randomized controlled trial in a primary care setting including 86 patients with stable HFpEF. Patients will undergo 3 study visits (a screening visit, a baseline visit and a post-intervention visit) including measurements of disease-specific biomarkers (using blood samples), cardiac and arterial vessel structure and function (using electrocardiogram, echocardiography, pulse wave velocity, flow-mediated dilation, retinal vessel analysis, cold pressure test), exercise tolerance (using spiroergometry), muscle function (using near-infrared spectroscopy, muscle strength tests), habitual physical activity (using accelerometry) and QoL. After the baseline visit, patients will be randomized to either the intervention or control group. The intervention group (n=43) will attend a supervised 12-week HIT on a bicycle ergometer, while the control group (n=43) will attend a supervised 12-week moderate-intensity continuous training (MCT). After 12 weeks, the study measurements will be repeated in all patients (intervention and control group) in order to monitor the effects of the intervention (post-intervention visit). At 6 months, 1, 2 and 3 years after the last study visit, telephone interviews will be performed to assess medical outcomes and QoL.

Outlook: This study is expected to add important knowledge about the potential utility of a novel treatment strategy in HFpEF patients, which may help to improve both, QoL and functional status. Moreover, the analysed biomarkers might be able to provide further insight into prognosis and pathogenesis of HFpEF.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent as documented by the patient's signature
* NYHA functional classes II-III
* Signs and symptoms of chronic HF:

  * Dyspnea, paroxysmal nocturnal dyspnea
  * Reduced exercise capacity, extended recovery after exercising
  * Fatigue
  * Peripheral edema (lower leg, ankle)
* EF (Ejection fraction) >50%
* Structural or functional changes in echocardiography:

  * LAVI (left atrial volume index) >34 ml/m2 OR
  * LVMI (left ventricular mass index) >115 g/m2 (men), >95 g/m2 (women) OR
  * E/E' (ratio between mitral peak velocity of early filling (E) to early diastolic mitral annular velocity (E')) >13 AND mean E' septal and lateral wall <9 cm/s
* NT-proBNP >125 pg/ml
* At least 4 weeks on stable medical treatment or without signs and symptoms of cardiac decompensation
* Trainable: Ventilatory threshold >40% of predicted VO2max AND VO2peak >10 ml/kg/min at the screening visit

Exclusion Criteria:

* Planned cardiac interventions in the following 6 months
* Unstable angina pectoris
* Paroxysmal atrial fibrillation
* Severe uncorrected valvular heart disease
* Uncontrolled brady- or tachyarrhythmia and hypertonic blood pressure
* Clinically significant concomitant disease states (e.g. advanced renal failure, hepatic dysfunction, insulin-dependent diabetes, COPD (chronic obstructive pulmonary disease) in grades III-IV, on-going cancer treatment)
* Significant musculoskeletal disease limiting exercise tolerance
* Active infection
* Immunosuppressive medical therapy
* Earlier hypersensitivity to parenteral iron preparation
* Anemia and iron deficiency due to active and/or chronic bleeding
* Blood transfusion within the previous 30 days
* Vulnerable persons (age <18 years, pregnant and breastfeeding women)
* Known or suspected non-compliance, drug or alcohol abuse
* Inability to follow the study procedures due to insufficient language skills, psychological disorders, dementia, etc.
* Participation in another intervention study
* Life-expectancy <6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2023-03 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Change in peak oxygen uptake (VO2peak) due to training | Baseline and 12 weeks
  VO2peak will be measured by spiroergometry at the baseline and post-intervention visit: an incremental symptom-limited exercise test on an electronically operated bicycle ergometer (eBike, General Electric Company, Fairfield, Connecticut, USA) using a fixed ramp protocol (start at 10 watts, increase of 10 watts/minute) will be conducted. The test will be performed in an air-conditioned laboratory in the early afternoon under non-fasting conditions. After a 2-minute warm-up at 10 watts, patients will be instructed to pedal at a constant rate of 60 rpm to exhaustion or until signs of ischemia or serious cardiac arrhythmias appear. The exercise bout will be followed by a cool-down at 25 watts for 10 minutes or until HR is dropping down below 100 beats/minute. VO2peak will be defined as the highest value reached during exercise.

SECONDARY OUTCOMES:
Change in disease-specific biomarkers | Baseline and 12 weeks
  Biomarkers such as NT-proBNP, Renin, AT-2, UCN-2, Osteopontin, sST2, Gal-3, GDF-15, Copeptin, Big-Endothelin-1, PlGF/sFlt-1, hs-CRP, IL-6 and IGF-BP7 will be measured. Furthermore, biomarkers for endothelial integrity, circulating mature endothelial cells and immature endothelial progenitor cells, systemic oxidative stress level and sarcopenia (irisin) will be assessed. Venous blood samples will be collected in serum or EDTA coated tubes (in total ~70ml). For serum isolation blood will be centrifuged and the serum will be frozen at -80°C and stored in the laboratory of the DSBG until the last participant will have completed the study procedures. Biomarkers except NT-proBNP will be analysed in external specialized laboratories or by trained personnel of the DSBG, if necessary. Whole blood will be immediately used to investigate circulating immature and mature endothelial progenitor cell numbers by flow cytometry - remaining mononuclear cells will be frozen at -80°C.
Change in echocardiographic parameters of the left ventricular systolic and diastolic function | Baseline and 12 weeks
  An echocardiography will be performed using a Full HD Color Doppler Ultrasound Scanner UF-890AG (Fukuda Denshi, Tokyo, Japan) by experienced echocardiographers blinded to the assignment of the patient to the intervention or control group, and independently analysed by trained study personal.
Change in arteriovenous oxygen difference (Da-vO2) | Baseline and 12 weeks
  Da-vO2 will be calculated using the Fick Principle: Peak Da-vO2 = VO2peak / peak cardiac output. VO2peak will be measured by spiroergometry, while peak cardiac output will be determined using the Full HD Color Doppler Ultrasound Scanner UF-890AG (Fukuda Denshi, Tokyo, Japan).
Change in pulse wave velocity (PWV) | Baseline and 12 weeks
  PWV will be measured at the same time as the echocardiographic parameters with the VaSera VS-2000 Vascular Screening System (Fukuda Denshi Co. Ltd, Tokyo, Japan) and evaluated by experienced blinded members of the study team.
Change in daily physical activity | Baseline and 12 weeks
  The number of daily steps, physical activity level and time spent at different walking speeds will be measured by the AiperMotion 440 PC (Aipermon GmbH, Munich, Germany), a three-axis accelerometer that is attached to the belt on the left hip, on 7 consecutive days for at least 12 hours a day with the exception of the time spent for showering, bathing and sleeping. For recording daily activities and non-wearing periods, patients will be asked to keep a diary.
Change in NYHA functional class | Baseline and 12 weeks
  NYHA functional class will be determined according to the New York Heart Association classification.
Change in quality of life (QoL): The 36-Item Short Form Health Survey (SF-36) | Baseline and 12 weeks
  The SF-36 consists of 36 items, which are formatted as binary questions or as semantic 6-point differential scales. It refers to the past 4 weeks and includes 9 content areas concerning vitality, general health perception, physical functioning, social functioning, role limitations (emotional/physical problems), pain, mental health and health change.
Change QoL: The Kansas City Cardiomyopathy Questionnaire (KCCQ) | Baseline and 12 weeks
  The KCCQ consists of 15 items concerning overall symptoms, emotional, social and mental status within the past 2 weeks.
Change in QoL: The Minnesota Living With Heart Failure Questionnaire (MLWHFQ) | Baseline and 12 weeks
  The MLWHFQ refers to the past 4 weeks and includes 21 questions on a 6-point scale with a maximum of 105 points (<24 good QoL, >45 poor QoL).
Change in body composition: Body Mass Index (BMI) | Baseline and 12 weeks
  BMI will be calculated from measured height in meters and weight in kilograms. Weight and height will be combined to report BMI in kg/m^2.
Change in body composition: Waist-to-Hip-Ratio (WHR) | Baseline and 12 weeks
  WHR will be calculated from measured waist circumference (WC) and hip circumference (HC) in centimetres. WC will be divided by HC to report WHR.
Change in macrovascular function: flow-mediated dilation (FMD) | Baseline and 12 weeks
  The flow mediated dilation (FMD) is a principle to measure the integrity of the endothelia. It refers to dilation of an artery when blood flow increases in that artery. The primary cause of FMD is release of nitric oxide by endothelial cells through shear stress. Flow-mediated dilatation (FMD) of the brachial arteries provides a non-invasive alternative to other measurement procedures. To determine FMD, brachial artery dilation following a transient period of forearm ischemia is measured using ultrasound (UNEFEX 38G 3.0, UNEX Co., Nagoya, Japan). The rationale behind the measurement is that endothelial cells are sentinels of cardiovascular health. Their function is reduced by the presence of cardiovascular risk factors, and is regained once pathological stimuli are removed
Change in microvascular function: retinal vessel analysis | Baseline and 12 weeks
  Static and dynamic retinal vessel analysis will be performed using the retinal vessel analysis system (RVA; IMEDOS Systems, Jena, Germany) and a fundus camera (450 FF; Carl Zeiss, Jena, Germany). We will take three valid images and two videos of the eye background to quantify retinal microvascular function. Conventional eye drops (Tropicamide 0.5%) will be used for pupil dilation of one eye, which is necessary for these measurements. All participants are asked to use public transport because of their dilated pupil. We recommend not to take part in road traffic for four hours after pupil dilatation. After this time, the vision should be normal again. In the first seconds after application of Tropicamide a light and temporary burning irritation or light headache are possible.
Change in macrovascular function: carotid artery reactivity | Baseline and 12 weeks
  Carotid artery reactivity (CAR) is a parameter, assessed noninvasively by transcutaneous ultrasound to examine endothelial function following sympathetic stimulation produced by the cold pressor test (CPT). Right carotid artery diameter is recorded before and during 90 seconds of immersion of the hand up to the wrist in ice water (4°C). Images will be obtained using a high-resolution ultrasound machine (UF-760AG, 5-12 MHz linear array transducer, Fukuda Denshi Co. Ltd., Tokyo, Japan).
Change in cardiovascular function: cardiac output | Baseline and 12 weeks
  The measurement of cardiac output will be performed with Cardioimpedanz (Physioflow, Manatec Biomedical, Poissy, France).
Change in muscular function: muscle oxygen saturation | Baseline and 12 weeks
  Muscle oxygen saturation is measured with Near infrared spectroscopy (NIRS, Portamon, Artinis Medical Systems, Elst, The Netherlands). NIRS relies mainly on two characteristics of human tissue. First, the relative transparency of tissue to light in the NIR range, and second, the oxygenation-dependent light absorbing characteristics of hemoglobin. By using a number of different wavelengths, the relative changes in hemoglobin concentration can be displayed continuously and saturation respectively absorption can be measured. If the absorption is known, the Lambert-Beer law can be used to calculate the chromophore's absorption. The technique on which NIRS relies is closely analogous to the technique of pulse oximetry and is in consequence not painful and not invasive.
Change in muscular function: muscle strength | Baseline and 12 weeks
  The strength test is a so-called Mid-Thigh-Pull Test. This isometric test is conceptualized in order to rate whole body force. The force of all extensors of the leg e.g. M. rectus femoris and of the back such as M. erector spinae as well as muscles of the hand. The test is comparable to elevate a table by hand. Two factors will be measured: the ability of a patient to generate maximum force ('Peak Force') and the second factor is measuring the increase of force over time (Rate of Force Development).

CONTACTS AND LOCATIONS:
Overall Officials: Arno Schmidt-Trucksäss, MD, Principal Investigator — University of Basel; Thomas Dieterle, MD, Principal Investigator — University of Basel
Locations (1):
- Department for Sport, Exercise and Health, Section Sports and Exercise Medicine, University of Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Patient-level anonymised datasets can be requested after completion of all planned analyses and publications from the study centre (anticipated by mid 2022). Public access to the study protocol will be granted by publishing it in a scientific journal. Blood sample results will be shared on the Swiss Biobanking Platform.

REFERENCES:
- [Derived] Gasser BA, Boesing M, Schoch R, Brighenti-Zogg S, Kropfl JM, Thesenvitz E, Hanssen H, Leuppi JD, Schmidt-Trucksass A, Dieterle T. High-Intensity Interval Training for Heart Failure Patients With Preserved Ejection Fraction (HIT-HF)-Rational and Design of a Prospective, Randomized, Controlled Trial. Front Physiol. 2021 Sep 24;12:734111. doi: 10.3389/fphys.2021.734111. eCollection 2021. PMID 34630155